CLINICAL TRIAL: NCT06774560
Title: Clinical Evaluation of 3D Printed Versus CAD/CAM Milled Onlays Over a Period of One Year: a Randomized Clinical Trial
Brief Title: Clinical Evaluation of 3D Printed Versus CAD/CAM Milled Onlays
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Sameh Ahmed Farouk, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3DP_CAD/CAMM
Record Dates: First submitted 2024-12-28; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Badly Decayed Molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAD/CAM milled onlays (Active Comparator): CAD/CAM has had a lasting impact on the dental market for decades. Its clinical reliability compared to any other dental material has been well documented. Several clinical studies proved its high clinical performance and survival rate. As CAD/CAM systems have become established in producing indirect restorations, it is considered the gold standard of digital manufacturing technology in dentistry.
  Interventions: Other: CAD/Cam milled onlays
- 3D printed onlays (Experimental): 3D-printed restorations have shown several advantages. Some studies have shown that the edge and internal gap values of 3D printing restorations are significantly lower than those of milling restorations.
  Interventions: Other: 3D printed onlays

INTERVENTIONS:
Other: CAD/Cam milled onlays — The digital workflow in dentistry has proven in the past decades to be a time-efficient, multifunctional, effortless, and accessible approach. The inherited shortages milling machines represented by the incapability to produce accurate complex hollow structures may give preference to modern 3D ceramic printing.
  Computer-aided-design/computer-aided-manufacturing (CAD/CAM) in dentistry is a digital subtractive approach for manufacturing indirect restorations. Nevertheless, waste materials and milling burs wearing are considered as key disadvantages of CAD/CAM technology, and are the main drive to improve 3D printing technology (additive manufacturing) as the latter has shown considerable efficiency in minimising wasted materials.
  Arms: CAD/CAM milled onlays
Other: 3D printed onlays — 3D printing technologies are developing more intensively in dentistry as this technology has the capacity to produce shapes or models with high accuracy and in a short time. This method of fabrication takes less time and money and saves on materials compared to CAD/CAM.
  Although it seems that digital manufacturing technology has made great changes in the restorative dentistry field, this technology is still not fully in use. This is possibly because of the lack of studies and research on this technology, particularly in terms of clinical performance and patient-centred outcomes. 3D printing technologies are novel technologies with a lack of research; therefore, the processing of 3D printing materials is still controversial.
  Arms: 3D printed onlays

SUMMARY:
The digital workflow in dentistry has proven in the past decades to be a time-efficient, multifunctional, effortless, and accessible approach. The inherited shortages milling machines represented by the incapability to produce accurate complex hollow structures may give preference to modern 3D ceramic printing.

Computer-aided-design/computer-aided-manufacturing (CAD/CAM) in dentistry is a digital subtractive approach for manufacturing indirect restorations. Nevertheless, waste materials and milling burs wearing are considered as key disadvantages of CAD/CAM technology, and are the main drive to improve 3D printing technology (additive manufacturing) as the latter has shown considerable efficiency in minimising wasted materials.

Although additive manufacturing has been known since the 1980s, its application in dentistry is relatively new and not fully studied with limited research and in vivo studies on their clinical performance.

ELIGIBILITY:
Inclusion Criteria:

Age: 25-45 years.

* Males or females.
* Participants with carious vital ower molars indicated for onlay (one or two missing cusps)
* Patients with at least 20 teeth under occlusion.
* Good oral hygiene.
* Co-operative patients approving to participate in the trial.
* Have sufficient cognitive ability to understand consent procedures.

Exclusion Criteria:

* Participants with parafunctional habits or bruxism.
* Participants with systemic diseases or disabilities that may affect participation.
* Heavy smoking.
* Pregnancy.
* Lack of compliance.
* Severe or active periodontal disease.
* Cognitive impairment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Fracture | One Year
  This outcome will be measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable, Charlie is not accepted

SECONDARY OUTCOMES:
Retention | One Year
  This outcome will be measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable, Charlie is not accepted
Marginal adaptation | One Year
  This outcome will be measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable, Charlie is not accepted
Marginal discoloration | One Year
  This outcome will be measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable, Charlie is not accepted
Secondary caries | One Year
  This outcome will be measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable, Charlie is not accepted
Post-operative hypersensitivity | One Year
  This outcome will be measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable, Charlie is not accepted
Surface texture | One Year
  This outcome will be measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable, Charlie is not accepted
Anatomic form | One Year
  This outcome will be measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable, Charlie is not accepted